CLINICAL TRIAL: NCT04626063
Title: The Effect of Magnesium Oral Supplementation for Acute Non-specific Low Back Pain: Prospective Randomized Clinical Trial
Brief Title: Magnesium Oral Supplementation for Acute Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Serkan Bayram, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/1330
Record Dates: First submitted 2020-11-01; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Low Back Pain; Acute Pain
MeSH Terms: conditions — Low Back Pain; Acute Pain | interventions — Magnesium; Anti-Inflammatory Agents, Non-Steroidal; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isolated non-steroid anti-inflammatory drug group (Active Comparator): A isolated NSAIDs group received 400 mg etodolac twice a day for 10 days in treatment of acute low back pain.
  Interventions: Drug: NSAID
- Non-steroid anti-inflammatory drug plus magnesium group (Experimental): This group received 400 mg etodolac twice a day and 365 mg magnesium oral supplementation once a day for 10 days in treatment of acute low back pain.
  Interventions: Drug: Magnesium
- Non-steroid anti-inflammatory drug plus paracetamol group. (Active Comparator): This group 400 mg etodolac twice a day and 500 mg paracetamol twice a day for 10 days in treatment of acute low back pain.
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: Magnesium — Patients were treated with etodolac 400mg twice a day plus magnesium oral supplementation once a day for acute low back pain and clinical evaluation of participants was performed at first admission to emergency department, at 4th and 10th days after the initiation of designated treatment
  Other Names: NSAID plus magnesium group
  Arms: Non-steroid anti-inflammatory drug plus magnesium group
Drug: NSAID — Patients were treated with etodolac 400mg twice a day for acute low back pain and and clinical evaluation of participants was performed at first admission to emergency department, at 4th and 10th days after the initiation of designated treatment
  Other Names: Isolated non-steroid anti-inflammatory group
  Arms: Isolated non-steroid anti-inflammatory drug group
Drug: paracetamol — Patients were treated with etodolac 400mg twice a day plus 500mg paracetamol twice a day paracetamol for acute low back pain and and clinical evaluation of participants was performed at first admission to emergency department, at 4th and 10th days after the initiation of designated treatment
  Other Names: NSAID plus paracetamol group
  Arms: Non-steroid anti-inflammatory drug plus paracetamol group.

SUMMARY:
Acute non-specific low back pain (LBP) is one of the most common complaints at the emergency department. It is more prevalent in countries with high-income economies, where 60-80% of the population report back pain at some point in their life. Numerous medication options are available for acute LBP relief such as non-steroid anti-inflammatory drugs (NSAIDs), myorelaxant drugs, opioids, and benzodiazepines. Magnesium is a physiological voltage-dependent blocker of N-methyl-D-aspartate NMDA)-coupled channels that can influence inflammatory pain and neuropathic pain through several different mechanisms. In this study the investigators aimed to investigate the effect of magnesium oral supplementation for acute low back pain.

DETAILED DESCRIPTION:
This study was conducted at our emergency department between June 2018 and March 2020 after receiving approval from our institutions' ethics committee (2018/1330). This study was registered as a randomized controlled trial with the US National Institute of Health (clinical trials.gov). We conducted a three-arm, prospective randomized open label clinical trial to compare isolated NSAID group, NSAID with paracetamol group and NSAID with oral magnesium supplementation group (described below) for treatment of acute LBP. Patients were included after providing informed consent predicated on their understanding of expected complications and treatment outcomes. Consolidate Standards of Reporting Trials (CONSORT) guidelines were followed reporting the results of the study Patients from a single university hospital were recruited for this study between June 2018 and March 2020. Inclusion criteria were defined as (1) age>18 years old, (2) duration of symptoms <2 weeks and (3) functionally impairing LBP which we defined as a score of > 5 on Roland-Morris Disability Questionnaire (RMDQ).

Exclusion criteria included (1) age>65 years old, (2) history of trauma, (3) presence of radicular pain physical examination which was defined as pain radiating below the gluteal folds, (4) history of primary vertebral tumor or metastasis, (4) patients who were pregnant or lactating, (5) presence of any contraindication or allergy to investigational medications, (6) history of chronic analgesic use, (7) history of autoimmune diseases or inflammatory rheumatic disorders, (8) history of cardiopulmonary restrictions, severe kidney or liver function disorders and (9) history of prior surgery of lumbar spine.

We based our sample size calculation assumptions on a recently published clinical trial [11] and widely accepted minimum clinically important improvement of 5 points on the RMDQ.(14) With alpha and beta values were set at 0.05 and 0.20 respectively, sample size calculation revealed that 50 patients were needed in each study group. To account for protocol violations, lost-to-follow-up and to ensure sufficient power for the intention to treat analysis (in previous work, up to 1/3 of enrolled patients did not use the investigational medication), we enrolled 80 patients for each group.

A computer generated random list was established with an online sequencer (www.random.org/sequences) according to which participants were randomly assigned to one of three study groups with 1:1:1 allocation ratio. Group A included isolated NSAID treatment and received 400 mg etodolac twice a day. Group B included NSAID and magnesium treatment and received a combination of 400 mg etodolac twice a day with 365 mg oral magnesium supplementation once a day. Group C included NSAID and paracetamol treatment and combination of 400 mg etodolac twice a day with 500 mg paracetamol twice a day was administered to the participants of this group (Figure-1). We effort to prevent the placebo effect by comparing the NSAID + magnesium therapy with both a NSAID plus paracetamol therapy and an isolated NSAID therapy. Treatment was performed by two authors (S.B and K.Ş) and patients were followed-up by same authors throughout the study. External medication was not allowed with the exception of topical analgesics. Patients who received any intravenous or intramuscular analgesia during the treatment period were excluded from study. Co-medications for any accompanying chronic condition (diabetes, hypertension etc.) were unchanged.

Clinical evaluation of participants was performed at first admission to emergency department, at 4th and 10th days after the initiation of designated treatment. Outcome measures included pain, mobility of lumbar spine and functional outcome. Pain intensity was assessed using a visual analogue scale (VAS). Lumbar spine mobility was assessed using the "finger to floor" test. Participants were asked to stand on erect posture with knees extended and then to bend forward in an attempt to reach for the floor with their fingertips without losing knee extension. Distance between patient's fingertips and the floor was then measured with a measuring tape. Functional outcome was evaluated with Roland-Morris Disability Questionnaire (RMDQ) score. RMDQ is a 24-item LBP functional scale and is recommended for research purposes. Higher scores signify greater low back-related functional impairment. An improvement of 5 points was considered clinically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients aged>18 years old,
* initiation of acute low back pain in the 10 days prior to study entry and functionally impairing low back pain, which we defined as a score of > 5 on the Roland-Morris Disability Questionnaire (RMDQ).

Exclusion Criteria:

* aged>65 years old,
* history of trauma,
* radicular pain, which we defined as pain radiating below the gluteal folds,
* history of vertebral tumor or metastasis,
* patients who were pregnant or lactating,
* unavailable for follow-up,
* with allergy or contraindication to the investigational medications,
* chronic analgesic use,
* autoimmune diseases or inflammatory rheumatic disorders,
* cardiopulmonary restrictions,
* severe kidney or liver function disorders and prior surgery on the lumbar spine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2020-03-08 (Actual)

PRIMARY OUTCOMES:
Changed of Baseline Roland-Morris Disability Questionnaire score at 10 days | Baseline, at 4th and 10th days
  This scoring system is consist of a 24-item low back pain functional scale recommended for use in low back pain research. Its yes/no format is amenable to telephone follow-up. Higher scores signify greater low back-related functional impairment.
Changed of Baseline VAS score at 10 days | Baseline, at 4th and 10th days
  Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10).

SECONDARY OUTCOMES:
Changed of Baseline Finger to floor test at 10 days | Baseline, at 4th and 10th days
  This test assess the mobility of lumbar spine. When test applied physical therapist say the patient to bend forward and attempt to reach for the floor with their fingertips. The physical therapist then measures the distance between the patient's right long finger and the floor using a standard measuring tape.

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Akgül, MD, Study Director — Istanbul University
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)